CLINICAL TRIAL: NCT02603705
Title: An Open-label Phase 3 Trial to Evaluate the Safety and Tolerability of Egalet ADER Oxycodone Tablet, Egalet-002, in Patients With Moderate-to-Severe Chronic Noncancer Pain
Brief Title: Safety and Tolerability of Egalet-002 in Patients With Moderate-to-Severe Chronic Noncancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-EG-303
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Moderate-to-severe Chronic Noncancer Pain
Keywords: chronic pain; opioid; oxycodone; non cancer pain; moderate to severe
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone extended-release (Experimental): Egalet abuse-deterrent, extended-release oxycodone tablet
  Interventions: Drug: Oxycodone extended-release

INTERVENTIONS:
Drug: Oxycodone extended-release

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Egalet-002 in opioid-experienced patients with moderate-to-severe chronic noncancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Is a man or woman between 18 and 75 years of age.
* Has a clinical history of moderate-to-severe chronic noncancer pain ≥6 months.
* Has required opioid therapy for at least 14 days prior to Screening at a dose between 20 mg and 160 mg (inclusive) oxycodone/day (or opioid equivalent), and will, in the opinion of the investigator, continue to require opioid therapy (between 20 mg and 240 mg oxycodone/day, inclusive) for management of moderate-to-severe pain for the duration of the study.
* Has pain either not adequately controlled on current opioid regimen, requires a change of opioid due to tolerability of current opioid regimen or in the opinion of the investigator, would benefit from changing opioid for another reason.
* Has stable health, as determined by the investigator.
* If female, the patient is currently not pregnant, not breast-feeding, nor attempting to become pregnant (for 30 days before screening through the duration of the study), or is of non-childbearing potential.
* Other Criteria Apply

Exclusion Criteria:

* Has cancer-related pain.
* Is receiving >240 mg oxycodone daily (or opioid equivalent) within 30 days before Screening.
* Has a history of attempted suicide.
* Has used a spinal infusion pump within 6 months before Screening.
* Has clinically unstable cardiac disease (including atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia) and/or respiratory disease (including chronic obstructive pulmonary disease or sleep apnea).
* Has positive urine toxicity screen for drugs of abuse (with the exception of prescribed medications).
* Has positive result for tetrahydrocannabinol (even if legally prescribed).
* Has current (or history of within the last 12 months) drug dependence or substance abuse disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, Text Revision criteria (excluding nicotine).
* Other Criteria Apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs during the Open-label Treatment Period, including those leading to treatment withdrawal, and/or abnormal physical examination findings, vital signs measurements, ECGs, and clinical laboratory test results, related to treatment | 1 year

SECONDARY OUTCOMES:
Findings of the Brief Pain Inventory-Short Form (BPI-SF) during the Open-label Treatment Period | 1 year

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Site 334, Huntsville, Alabama
  - Site 328, Tucson, Arizona
  - Site 332, Jacksonville, Florida
  - Site 340, Miami Gardens, Florida
  - Site 320, Plantation, Florida
  - Site 302, Tampa, Florida
  - Site 315, Tampa, Florida
  - Site 310, Winter Haven, Florida
  - Site 316, Dawsonville, Georgia
  - Site 311, Marietta, Georgia
  - Site 336, Bloomington, Illinois
  - Site 345, Blue Island, Illinois
  - Site 304, Evansville, Indiana
  - Site 325, Valparaiso, Indiana
  - Site 321, Overland Park, Kansas
  - Site 342, Wichita, Kansas
  - Site 329, New Orleans, Louisiana
  - Site 326, Quincy, Massachusetts
  - Site 303, St Louis, Missouri
  - Site 306, Las Vegas, Nevada
  - Site 313, Belvidere, New Jersey
  - Site 346, Blackwood, New Jersey
  - Site 323, Hartsdale, New York
  - Site 338, Mooresville, North Carolina
  - Site 333, Cincinnati, Ohio
  - Site 343, Cleveland, Ohio
  - Site 308, Huber Heights, Ohio
  - Site 347, Kettering, Ohio
  - Site 335, Oklahoma City, Oklahoma
  - Site 312, Eugene, Oregon
  - Site 322, Duncansville, Pennsylvania
  - Site 324, Wyomissing, Pennsylvania
  - Site 344, Myrtle Beach, South Carolina
  - Site 314, Summerville, South Carolina
  - Site 341, New Tazewell, Tennessee
  - Site 318, Austin, Texas
  - Site 330, Dallas, Texas
  - Site 309, San Antonio, Texas
  - Site 331, West Jordan, Utah